CLINICAL TRIAL: NCT02553811
Title: Accuracy of Ultrasonography and Electromyography in the Diagnosis of Carpal Tunnel Syndrome
Brief Title: Diagnosis of Carpal Tunnel Syndrome: Effectiveness of Diagnostic Tests. Clinical Trial of Accuracy
Acronym: DCTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Benedito Felipe Rabay Pimentel, master, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 244468
Record Dates: First submitted 2015-09-10; First posted 2015-09-18 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Carpal Tunnel Syndrome; Compression Neuropathy, Carpal Tunnel; Median Neuropathy, Carpal Tunnel
Keywords: carpal tunnel syndrome; clinical examination; diagnosis; clinical trial; median nerve compression; accuracy; ultrasonography; electromyography; electrodiagnostic testing
MeSH Terms: conditions — Carpal Tunnel Syndrome; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): accuracy diagnostic in carpal tunnel syndrome = evaluation and comparison ultrasonography X electromyography
  Interventions: Diagnostic Test: accuracy diagnostic

INTERVENTIONS:
Diagnostic Test: accuracy diagnostic — effectiveness of the ultrasonography and electromiography for best performance and diagnostic accuracy in carpal tunnel syndrome
  Other Names: accuracy of the ultrasonography; accuracy of the electromiography

SUMMARY:
There is no golden universal standard for the diagnosis of Carpal Tunnel Syndrome (CTS). In this scenario, for a comparison of the effectiveness of the principal diagnostic tests CTS should determine how they affect the likelihood of disease through a clinical accuracy trial of good methodological quality in order to get answers to what is the best diagnostic strategy in clinical CTS practice. The paresthesia in nerve distribution territory median hands is the most common symptom in patients with CTS. The nuisance caused by paresthesia directly affects the quality of life of patients and impairs daily manual activities and sleep quality. To evaluate the remission of paresthesia is a major clinical criterion for improved STC being an expected relevant outcome for the patient. This study evaluated and compared the diagnostic accuracy of the ultrasonography (US) and electromyography (EMG), considering the postoperative status of remission of paresthesia as the reference standard in the diagnosis of CTS.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is characterized by median nerve compression at the level of the wrist. It represents 90% of compressive neuropathies and is the most common upper member. For being a major cause of disability in hands, the early and accurate diagnosis to obtain a definitive treatment in CTS is essential. Despite this, there is no consensus on which is the most effective diagnostic criteria for CTS. The absence of a reference standard universally accepted for the diagnosis of CTS contributes to this scenario.

Ultrasonography (US) and electromyography (EMG) are the complementary examinations most often used in the diagnosis of CTS, but overestimated in their performance and require caution in interpreting the results, particularly the lack of a consensus on the ideal cutoff point for considering the diagnosis of CTS. This results in a wide variation in results of sensitivity and specificity for these tests, both the EMG (sensitivity = 82 to 98% and specificity = 19 to 88%) and for the US (sensitivity = 70 to 98% and specificity = 63 to 100%), in addition to a high proportion (20-40%) of false-negative and false-positive.

Most diagnostic accuracy studies at CTS compare the results of the US with EMG, considering most of the time the EMG as reference standard. There are few studies comparing the results of the US and EMG using other benchmarks, such as the degree of clinical improvement after surgical treatment of CTS or a combination of clinical signs and symptoms. The value of diagnostic tests for CTS can be established by comparing the diagnostic strategies and studying how they can affect the likelihood of STC. This spectrum can be considered the results of surgical treatment as the reference standard, as these are directly related to the diagnosis of CTS. Surgical treatment by classical open surgery is the definitive treatment of CTS and provides relief from symptoms, mainly the remission of paresthesia, with satisfactory results in up to 98% of the cases. The discomfort caused by paresthesia in the quality of life of patients and impairs daily manual activities and the quality of sleep is considerable in CTS. The remission of paresthesia is a clinical improvement parameter of the disease being an expected and relevant outcome for the patient. Primary and well-designed controlled studies with good methodological quality to guide the diagnostic practices and evaluate their effectiveness in an integrated manner in carpal tunnel syndrome (CTS) are unusual and challenging in the current literature. This study, innovative in its method has as primary objective to compare the accuracy of ultrasonography in relation electromyography in the diagnosis of carpal tunnel syndrome, using to the results of the surgical treatment as the reference standard.

The study design is a clinical trial of accuracy, primary, longitudinal, controlled, prospective, and performed in a single center. This clinical trial follows the accuracy STARD recommendations (Standards for Reporting of Diagnostic Accuracy).

Patients with clinical suspicion of CTS, who were referred and attended consecutively in our specialty clinic in hand surgery, were submitted to an initial clinical evaluation (ACI), by a same specialist in hand surgery, who used the CTS-6 clinical diagnostic instrument of GRAHAM et al. (2006), represented by a logistic regression model that estimates the diagnostic probability of CTS based on the presence or absence of the 6 diagnostic criteria that are: paresthesia, night paresthesia, weakness and/or atrophy thenar musculature, Tinel signal, Phalen test and loss of 2-points discrimination.

Diagnostic intervention of the US and EMG were performed by the same professional in each area, both experienced and specialized in their acting area, who were unaware of the clinical situation of patients at the time of the tests.

The ultrasonography (US) of the wrist were performed in a Philips brand equipment (model M2540A, Bothell, WA USA) with broadband linear transducers. The US examination technique consisted of the positioning of the patient comfortably, sitting with forearm in a supine position in slight flexion supported on the examination table, with the handle in neutral position and the hand with the fingers in extension. In order to assess the accuracy of the US in the diagnosis of CTS, a cutoff value equal to and greater than 10.0 mm² of the median nerve transverse cross-sectional area was considered at the proximal limit of the carpal tunnel.

The electromyography (EMG) of the upper limbs were performed on Nihon Kohden brand equipment (model MEB 9400K, 2 channels, Tokyo, Japan). The EMG technique consisted of the positioning of the patient comfortably, in a horizontal dorsal decubitus position with the head resting on a high headboard on the examination table and with the upper limbs positioned at rest along the body. The objective of the EMG was to determine the sensory conduction velocity of the median nerve in the third finger-cuff segment at a distance of 13 cm, with a cut-off value of less than 50 m/s and a higher value or equal to 4.2 ms for distal motor dormancy of the median nerve of the wrist to the tenar eminence (short abductor muscle of the thumb).

After the examinations of US and EMG, the patients were referred and submitted surgical treatment by classical open pathway, by a same surgeon. Outpatient surgeries were performed at the surgical center of the Vale do Paraíba Regional Hospital in Taubaté - SP. The anesthesia technique used was Bier's regional endovenous. Each patient was followed monthly until the fourth postoperative month.

To analyze the accuracy of the diagnostic tests of US and EMG in relation to the reference standard (remission of paresthesia), the McNemar test and the 2x2 contingency table were used, using as reference standard the improvement of paresthesia. The evolution of the Boston score by moments of evaluation and diagnostic results was evaluated using the analysis of variances (Anova) with repeated measures. Comparison of the means of the two groups was performed using the Student's t-test for independent samples. The analyzes were performed using the statistical package SPSS 20.0 and Stata 12. For all statistical tests, a significance level of 5% was adopted. The statistical sampling was performed considering a 20% difference between the sensitivity of the EMG and US diagnostic tests using the McNemar test, with a statistical power of 84.0% and a significance level of 5%. For this calculation, the value of 60% and a prevalence of 80% for STC were assumed as a percentage of total agreement, requiring a total sample of 115 patients. A further 5% of all patients were recruited to cover possible losses or exclusions during the course of the study. Statistical software PASS 14 (Power Analysis and Sample Size System) - NCSS was used.

There is a lack of accuracy of properly designed studies with good quality evidence to recommend good diagnostic practices in CTS. This study presents the innovative proposal of conducting a clinical trial of accuracy, specifically designed when there is no reference standard defined for the diagnosis of the CTS, using the reference paresthesia after surgery as a relevant outcome from the standpoint of the patient. The use of more accurate diagnostic criteria with a more effective diagnostic protocol for the clinical examination, the US and the EMG, based on a high level of evidence will lead directly into the paradigm shift for clinical decision-making, effective and safe CTS treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients with a CTS-6 clinical diagnostic instrument of GRAHAM et al. (2006) with score equal to or greater than 12 points
* Female gender
* Aged 40 to 80 years
* Patients with unilateral or bilateral involvement (only one hand was considered for inclusion)
* Patients who agreed to participate in this study and who signed the informed consent form (TCLE)
* Patients who underwent some kind of previous conservative treatment for CTS without clinical improvement.

Exclusion criteria:

* Cervical radiculopathy
* Thoracic outlet syndrome
* Pronator syndrome
* Patients with history of previous surgical release of the carpal tunnel
* Patients with sequelae of fracture of the wrist
* Patients who did not agree to participate or who did not sign the TCLE.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of the ultrasonography (US) | four months
  Patients with CTS who obtained as a result of surgical treatment, remission of paresthesia were considered to be truly ill, and patients who did not receive remission of paresthesia were considered non-diseased. The remission of paresthesia evaluated after surgical treatment was considered the reference standard for the diagnosis of CTS. The accuracy of US was assessed by evaluating the results of the US (positive or negative) in relation to the results of surgery (remission of paresthesia or non-remission of paresthesia).
Accuracy of the electromyograph (EMG) | fours months
  Patients with CTS who obtained as a result of surgical treatment, remission of paresthesia were considered to be truly ill, and patients who did not receive remission of paresthesia were considered non-diseased. The remission of paresthesia evaluated after surgical treatment was considered the reference standard for the diagnosis of CTS. The accuracy of EMG was assessed by evaluating the results of the EMG (positive or negative) in relation to the results of surgery (remission of paresthesia or non-remission of paresthesia).
Life quality | fours months
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a disease-specific STC questionnaire, self-administered, translated and validated for the Portuguese language, which evaluates two components: a symptom severity scale with 11 questions and a functional status scale with 8 issues. All patients in this study responded to two BCQT, the first after initial clinical evaluation and the second at the end of the fourth month of postoperative follow-up. To assess the improvement of severity and functional status of the patients in this study, a medically significant improvement in the two scales was expected between the means of the second Boston questionnaire (according to BCQT) compared to the means of the first Boston questionnaire (first BCQT).

SECONDARY OUTCOMES:
Improvement in severity of symptoms and functional status of the patients | four months
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a disease-specific STC questionnaire, self-administered, translated and validated for the Portuguese language, which evaluates two components: a symptom severity scale with 11 questions and a functional status scale with 8 issues. All patients in this study responded to two BCQT, the first after initial clinical evaluation and the second at the end of the fourth month of postoperative follow-up. To assess the improvement of severity and functional status of the patients in this study, a medically significant improvement in the two scales was expected between the means of the second Boston questionnaire (according to BCQT) compared to the means of the first Boston questionnaire (first BCQT).

CONTACTS AND LOCATIONS:
Overall Officials: João C Belloti, researcher, Principal Investigator — Federal University Of the São Paulo
Locations (1):
- Hospital Regional do Vale do Paraiba, Taubaté, São Paulo, Brazil

REFERENCES:
- [Result] Pimentel B F, Abicalaf C A, Braga L, Albertoni W M, Fernandes C H, Sernik R A, Faloppa F. Cros-sectional area of the median nerve characterized by ultrasound in patients with carpal tunnel syndrome before and after release of the transverse carpal ligament. Journal of Diagnostic Medical Sonography 2013; 29(3):116-121. Graham B, Regehr G, Naglie G, Wright J G. Development and validation of diagnostic criteria for carpal tunnel syndrome. J Hand Surg 2006; 31A: 919-924 D'Arcy C A, McGee S. The rational clinical examination. Does this patient have carpal tunnel syndrome ? JAMA 2000; 283(23): 3110-3117. McCabe S. Evidence-Based Medicine - Diagnosis of Carpal Tunnel Syndrome. J Hand Surg 2010; 35A: 646-648. Sernik R A, Abicalaf C A, Pimentel B F, Braga-Baiak A, Braga L, Cerri G G. Ultrasound features of carpal tunnel syndrome: a prospective case-control study. Skelectal Radiol 2008; 37: 49-53.
- [Derived] Pimentel BFR, Faloppa F, Tamaoki MJS, Belloti JC. Effectiveness of ultrasonography and nerve conduction studies in the diagnosing of carpal tunnel syndrome: clinical trial on accuracy. BMC Musculoskelet Disord. 2018 Apr 12;19(1):115. doi: 10.1186/s12891-018-2036-4. PMID 29649998